CLINICAL TRIAL: NCT00073372
Title: Abciximab (ReoPro) in Acute Ischemic Stroke: A Phase III, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: A Study of Effectiveness and Safety of Abciximab in Patients With Acute Ischemic Stroke (AbESTT-II)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on the data and observed benefit-risk profile, the trial's independent oversight committee recommended that enrollment not resume.
Sponsor: Centocor, Inc. (Industry)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004768
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-06

CONDITIONS: Cerebrovascular Accident; Brain Ischemia; Acute Disease
Keywords: Acute ischemic stroke; abciximab; ReoPro; drug safety; drug efficacy; intracranial hemorrhage; stroke
MeSH Terms: conditions — Stroke; Brain Ischemia; Acute Disease; Ischemic Stroke; Intracranial Hemorrhages | interventions — Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Abciximab

SUMMARY:
The purpose of this study is to determine the effectiveness of abciximab in the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
Abciximab is a drug that prevents platelets from sticking together and forming a clot. There are limited studies using abciximab in the treatment of strokes. This phase III, multicenter, randomized, double-blind, placebo-controlled, parallel group study is designed to assess the effectiveness and safety of abciximab for treatment of acute ischemic stroke, in helping dissolve clots in brain arteries so that blood and oxygen can flow better and there may be less brain damage.

Safety evaluations will be performed at specified intervals throughout the study and will consist of laboratory tests, vital signs (such as blood pressure), physical examinations and the occurrence and severity of adverse events as well as other study specific procedures. Patients will receive either Abciximab: 0.25 mg/kg bolus (to a maximum of 30 mg) followed by a 0.125 µg/kg/min infusion (to a maximum of 10 µg/min) for 12 hours or a bolus of placebo followed by infusion for 12 hours

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of acute ischemic stroke with onset within 5 hours and 30 minutes before randomization and planned treatment initiation within 6 hours of onset
* After 600 patients are enrolled in previous criteria, the new criteria for enrollment will be, patients with diagnosis of acute ischemic stroke with onset within 4 hours and 30 minutes before randomization and planned treatment initiation within 5 hours of onset

Exclusion Criteria:

* Patients who had participation in another study with an investigational drug or device within the last 30 days, prior participation in the present study, or planned participation in another trial
* Patients with symptoms suggestive of subarachnoid hemorrhage
* Female patients known to be pregnant, lactating, or having a positive or indeterminate pregnancy test
* Patients with neurological deficit that has led to stupor or coma
* Patients with minor stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2003-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The proportion of modified Rankin Scale responders at 3 months in the primary population.

SECONDARY OUTCOMES:
Proportion of patients with neurological recovery and all-cause mortality at 3 months in the primary population. Fatal intracranial-, nonfatal symptomatic parenchymal-, or other symptomatic intracranial hemorrhages though discharge at day 5 & 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Adams HP Jr, Effron MB, Torner J, Davalos A, Frayne J, Teal P, Leclerc J, Oemar B, Padgett L, Barnathan ES, Hacke W; AbESTT-II Investigators. Emergency administration of abciximab for treatment of patients with acute ischemic stroke: results of an international phase III trial: Abciximab in Emergency Treatment of Stroke Trial (AbESTT-II). Stroke. 2008 Jan;39(1):87-99. doi: 10.1161/STROKEAHA.106.476648. Epub 2007 Nov 21. PMID 18032739
- See also: Abciximab (ReoPro�) in Acute Ischemic Stroke: A Phase 3, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled Trial — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=146&filename=CR004768_CSR.pdf